CLINICAL TRIAL: NCT06454422
Title: Implementing the Wuqinxi on Patients With Pulmonary Arterial Hypertension to Enhance Exercise Tolerance ，Reduce Negative Emotions and Quality of Life: A Randomized Clinical Trial
Brief Title: Implementing the Wuqinxi on Patients With Pulmonary Arterial Hypertension
Acronym: PAH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: KY20240422-KS-01
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Arterial Hypertension PAH

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wuqinxi (Experimental): including observation of disease progression and complications, oxygen inhalation, medication guidance, rest and diet nursing, daily activity guidance, psychological guidance, and follow-up after discharge.
  Patients mimicked precise Wuqinxi movements and breathing patterns while exercising.
  Interventions: Other: wu qinxi
- general nursing routines (No Intervention): including observation of disease progression and complications, oxygen inhalation, medication guidance, rest and diet nursing, daily activity guidance, psychological guidance, and follow-up after discharge.

INTERVENTIONS:
Other: wu qinxi — Wuqinxi, also known as the Hundred-step Sweating Exercise, is one of the most emblematic Health qigong exercises. Huatuo, guided by the principle, formulated the 'Wuqinxi': " Running water is never stale and a door-hinge is never gets worm-eaten," and sums up the experiences of the fitness activities of Huatuo's predecessors that imitate the movements of tigers, deer, bears, apes, birds, and other animals, and are associated with human organs, meridians, and 'qi'
  Arms: Wuqinxi

SUMMARY:
Aims and objective: The primary objective of this study was to assess the effects of a traditional Chinese Qigong practice known as Wuqinxi on activity tolerance，negative emotions and quality of life in pulmonary arterial hypertension patients.

Methods: In the current prospective, randomized-controlled clinical trial, 60 patients with pulmonary arterial hypertension were randomly assigned to one of two groups: intervention or control. Participants in the intervention group received targeted pharmacological therapy and five sessions of qigong exercise per week. In contrast, individuals in the control group underwent targeted drug therapy and routine care. Observe the change in exercise tolerance as measured by the 6-minute walking distance (6MWD). Serological indicators (n-terminal brain natriuretic peptide precursor, NT-pro BNP) ,negative emotions(PHQ-9/GAD-7)and the MOS Item Short Form Health Survey (SF-36) or emPHasis-10 were used to assess patients condition and quality of life.

DETAILED DESCRIPTION:
In the previous study, we examined the effects of comprehensive respiratory function exercise on exercise tolerance in patients with PAH. The results indicated that limb exercise combined with breath regulating guidance affects patients' physical health.Given these TCM principles, the current study investigated the clinical utility of Wuqinxi for improving patients' exercise tolerance and quality of life by comparing the intervention and control groups' NT-pro BNP scores, 6MWD data, negative emotionsand quality of life indices.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients with PAH related to IPAH(idiopathic pulmonary arterial), CTD(connective tissue disease), DPAH(drug-induced pulmonary hypertension), CHD(congenital heart disease) and associated with secondary disease, aged 18-75 years; (2)patients with PAH as defined by the American College of Cardiology Foundation/American Heart Association (right heart catheterization: mPAP≥20mmHg and PAWP≤15mmHg); (3) patients with WHO pulmonary arterial hypertension functional class II-III; (4) patients on drug-based treatment for ≥1 month and in the recovery period; (5) could read, write, and comprehend Chinese; (6) volunteered for this trial and provided written informed consent.

Exclusion Criteria:

* (1) patients unable or unwilling to complete the 6MWD; (2) The physician confirms that the disease requires bed rest or with severely impaired cardiopulmonary function, tumors, and limb dysfunction; (3) patients who were unable to complete the questionnaire independently; (4) a history of mental problems and cognitive impairment; or have had psychotherapy or taken any psychiatric medication in the past or present.(5) patients who were hospitalized with severe disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Biomarker | admission and discharge at the end of 3 months
  NT-pro BNP was detected using a colloidal gold immunochromatography analyzer, model LEPU Quant 800, made in Beijing, China.
6-minute walking distance | admission and discharge at the end of 3 months
  The 6MWD test for selected patients with stable illness was conducted in the corridor of the cardiology ward
Quality of Life Assessment | admission and discharge at the end of 3 months
  emPHasis-10 or pulmonary hypertension health quality of life score, SF-36

SECONDARY OUTCOMES:
Negative emotions | admission and discharge at the end of 3 months
  PHQ-9/GAD-7

OTHER OUTCOMES:
Frail | admission and discharge at the end of 3 months
  Frail questionnaire
Nutrition | admission and discharge at the end of 3 months
  Simple Nutrition Assessment (MNA)
Sleep | admission and discharge at the end of 3 months
  Pittsburgh Sleep Quality Index (PSQI)

CONTACTS AND LOCATIONS:
Overall Officials: Chang yun, Study Chair — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No